CLINICAL TRIAL: NCT00742586
Title: Identification of Autonomic Failure Patients, Controls and Blood Sampling for Pilot Study
Brief Title: Autonomic Failure Patients for RNA Blood Sampling
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Western Michigan University (Other)
Responsible Party: Principal Investigator, David Robertson, Professor of Medicine, Pharmacology and Neurology, Vanderbilt University
Other Study IDs: 080373
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Pure Autonomic Failure; Multiple System Atrophy; Parkinson's Plus Syndromes
Keywords: Gene Expression Changes in Blood Cells; RNA; Pure Autonomic Failure; Multiply System Atrophy; Parkinson's Plus
MeSH Terms: conditions — Pure Autonomic Failure; Multiple System Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify 15 patients with autonomic failure and obtain blood samples for RNA from those participants and 15 control subjects within the same age range. The stabilized blood samples, along with a limited data set, will be shipped to Western Michigan University where the actual laboratory analysis (a separate study) of the samples will take place.

Unique genetic inscriptions, called gene expression signatures, are currently being identified for many diseases, including neurological diseases. The secondary goal of this study is to support the research being done at WMU and they try to look for MSA-specific signs are present in whole blood samples of MSA patients at late-stages of the disease. This is a pilot study that has a long term goal (through additional studies) a MSA-specific gene expression signature for the development of a diagnostic test for this disease that can be used in the future. Other patient groups with autonomic failure, characterized by significant drop in blood pressure on standing, will also be included in this study, to look for similar genetic inscriptions.

This pilot study is expected to last for 2 years. The investigators at WMU will need some de-identified health Information about the subjects, including their age at diagnosis, age (when sample drawn) and list of their medications

DETAILED DESCRIPTION:
Patients with one of the following autonomic problems will be recruited to participate in this study: multiple systems atrophy (MSA), pure autonomic failure (PAF) or Parkinson's Plus. The study consists of drawing 15 ml of whole blood for RNA. The blood is drawn in special collection tubes to stabilize the RNA material in the blood. The samples will be frozen and shipped to WMU for analysis.

The patients will also be asked to provide the current list of their medications, their age and the age when they were first diagnosed with their neurologic or autonomic disorder. This information will be de-identified and sent to the investigators at WMU as a limited data set.

ELIGIBILITY:
Inclusion Criteria for patients:

* presumed or probably diagnosis of autonomic disorder characterized by orthostatic hypotension
* age between 50 - 75 years
* Male or female
* Able and willing to provide consent

Inclusion Criteria for controls:

* Absence of neurological disorder
* age between 50 - 75 years
* Male or female
* Able and willing to provide consent

Exclusion Criteria:

* inability to provide consent

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 patients with diagnosis of autonomic disorder characterized by orthostatic hypotension, Pure Autonomic Failure, Multiple System Atrophy or Parkinson's Plus.
  15 controls without a neurological disorder
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Robertson, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States